CLINICAL TRIAL: NCT02757872
Title: Effects of Vitamin D and Fish Oil on the Kidney in Hypertensives
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Brigham and Women's Hospital (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2014-3778; R01DK102952 (NIH)
Record Dates: First submitted 2016-04-28; First posted 2016-05-02 (Estimated); Results first posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Hypertension; Kidney Diseases
Keywords: Hypertension; Kidney Diseases; Vitamin D; Omega 3 fatty acids
MeSH Terms: conditions — Hypertension; Kidney Diseases | interventions — Cholecalciferol; Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Intervention Model Description: Parent (VITAL; NCT01169259) study was based upon a 2x2 factorial design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin D and Omega-3 Fatty acids (Active Comparator): Dietary Supplement: Vitamin D Vitamin D3 (cholecalciferol), one 2000 IU capsule per day.
  Drug: Omega-3 fatty acids (fish oil) Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Interventions: Dietary Supplement: Vitamin D3; Drug: Omega-3 Fatty acids
- Vitamin D and Omega-3 Fatty acid Placebo (Active Comparator): Dietary Supplement: Vitamin D Vitamin D3 (cholecalciferol), one 2000 IU capsule per day.
  Dietary Supplement: Omega-3 fatty acid placebo (Fish oil placebo)
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Fish oil placebo
- Vitamin D Placebo and Omega-3 Fatty acids (Active Comparator): Drug: Omega-3 fatty acids (fish oil) Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Dietary Supplement: Vitamin D placebo. One capsule per day Vitamin D3 placebo
  Interventions: Drug: Omega-3 Fatty acids; Dietary Supplement: Vitamin D3 placebo
- Vitamin D Placebo and Omega-3 Fatty acid Placebo (Placebo Comparator): Dietary Supplement: Vitamin D placebo. One capsule per day Vitamin D3 placebo
  Dietary Supplement: Omega-3 Fatty acid Placebo (Fish oil placebo). One capsule per day
  Interventions: Dietary Supplement: Vitamin D3 placebo; Dietary Supplement: Fish oil placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D3 (cholecalciferol), 2000 IU per day
  Arms: Vitamin D and Omega-3 Fatty acid Placebo; Vitamin D and Omega-3 Fatty acids
Drug: Omega-3 Fatty acids — Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  Other Names: Fish oil
  Arms: Vitamin D Placebo and Omega-3 Fatty acids; Vitamin D and Omega-3 Fatty acids
Dietary Supplement: Vitamin D3 placebo — Vitamin D3 placebo
  Arms: Vitamin D Placebo and Omega-3 Fatty acid Placebo; Vitamin D Placebo and Omega-3 Fatty acids
Dietary Supplement: Fish oil placebo — Fish oil placebo
  Arms: Vitamin D Placebo and Omega-3 Fatty acid Placebo; Vitamin D and Omega-3 Fatty acid Placebo

SUMMARY:
The VITamin D and OmegA-3 TriaL (VITAL; NCT01169259) is an ongoing randomized clinical trial in 25,875 US men and women investigating whether taking dietary supplements of vitamin D3 (2000 IU) or omega-3 fatty acids (Omacor (R) fish oil, 1 gram) reduces the risk of developing cancer, heart disease, and stroke in people who do not have a prior history of these illnesses. The VITAL Kidney Function in Hypertension ancillary study will evaluate the effects of vitamin D or omega-3 fatty acids on kidney function among participants with baseline hypertension.

DETAILED DESCRIPTION:
This ancillary study to the VITamin D and OmegA-3 TriaL (VITAL) will test whether vitamin D3, omega-3 fatty acids, or both prevent the development and progression of kidney disease in participants with hypertension. Persons with hypertension are at high risk of kidney disease.

Vitamin D and omega-3 fatty acids are promising interventions for kidney disease prevention and treatment, based on results of animal-experimental models and early human studies. Because these interventions are relatively safe, inexpensive, and widely available, they may offer opportunity to substantially reduce the burden of kidney disease in large populations. This VITAL ancillary study will test whether vitamin D3 and/or omega-3 fatty acids prevent loss of glomerular filtration rate, over 4 years of therapy.

In VITAL, 25,875 participants have been randomly assigned in a 2x2 factorial design to vitamin D3 (cholecalciferol) 2000 IU daily versus placebo, and to eicosapentaenoic acid 465 mg plus docosahexaenoic acid 375 mg daily versus placebo, and followed for a mean of 5 years to assess effects on cardiovascular disease and cancer events. This ancillary study will identify and recruit a sub-cohort of VITAL participants with hypertension at baseline and ascertain effects of study interventions on glomerular filtration rate in this group. Blood samples will be collected at year 4 simultaneously for measurement of estimated glomerular filtration rate (using serum creatinine and cystatin C) and other relevant biomarkers. This VITAL ancillary study is designed to determine whether vitamin D3 and/or omega-3 fatty acids have causal and clinically relevant effects on the development and progression of kidney disease in hypertensives.

ELIGIBILITY:
Inclusion Criteria:

* Participants in VITAL (NCT01169259) with a self-reported physician diagnosis of hypertension are eligible to participate in this ancillary study

Exclusion Criteria:

* Diagnosis of diabetes mellitus

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2232 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michal L Melamed, MD, MHS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D Placebo and Omega-3 Fatty Acids Placebo: Dietary Supplement: Vitamin D placebo. One capsule per day Vitamin D3 placebo
  Dietary Supplement: Omega-3 Fatty acid Placebo (Fish oil placebo). One capsule per day
Period: Overall Study
Arm/Group | Vitamin D and Omega-3 Fatty Acids | Vitamin D and Omega-3 Fatty Acid Placebo | Vitamin D Placebo and Omega-3 Fatty Acids | Vitamin D Placebo and Omega-3 Fatty Acids Placebo
Started | 545 | 570 | 576 | 541
Completed | 545 | 570 | 576 | 541
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D and Omega-3 Fatty Acids | Vitamin D and Omega-3 Fatty Acid Placebo | Vitamin D Placebo and Omega-3 Fatty Acids | Vitamin D Placebo and Omega-3 Fatty Acids Placebo | Total
Number analyzed (Participants) | 545 | 570 | 576 | 541 | 2232
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (6.0) | 69.0 (6.4) | 69.0 (6.2) | 68.3 (6.1) | 68.7 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 278 | 309 | 303 | 285 | 1175
  Male | 267 | 261 | 273 | 256 | 1057
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 438 | 437 | 442 | 419 | 1736
  Non-Hispanic Black | 58 | 79 | 79 | 73 | 289
  Hispanic or Latino | 15 | 17 | 19 | 16 | 67
  Asian/Pacific Islander | 5 | 6 | 4 | 9 | 24
  American Indian or Alaskan Native | 3 | 5 | 4 | 5 | 17
  Other | 12 | 11 | 13 | 8 | 44
  Unknown | 14 | 15 | 15 | 11 | 55
Region of Enrollment [Number; unit: participants]
  United States | 545 | 570 | 576 | 541 | 2232
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.89 (0.23) | 0.89 (0.24) | 0.90 (0.35) | 0.87 (0.22) | 0.89 (0.26)

OUTCOME MEASURES:

1. Primary Outcome: Change in Estimated Glomerular Filtration Rate
Description: Serum creatinine and cystatin C measurement pre-randomization and year 4
Time Frame: Baseline and 4 years
Population: Glomerular filtration rate data was not collected as samples were never analyzed.
Arm/Group | Vitamin D and Omega-3 Fatty Acids | Vitamin D and Omega-3 Fatty Acid Placebo | Vitamin D Placebo and Omega-3 Fatty Acids | Vitamin D Placebo and Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Confirmation of Microalbuminuria
Description: Number of participants with positive Microalbuminuria was reported. Participants were defined as having positive microalbuminuria if their lab results were >30 mg/g Creatinine
Time Frame: 4 years post-randomization
Population: Urine samples were not collected from 34 participants in the 'Vitamin D and Fish Oil' group; 41 participants in the 'Vitamin D and Fish Oil Placebo' group; 33 participants in the 'Vitamin D Placebo and Fish Oil' group; and 35 participants in the 'Vitamin D Placebo and Fish Oil Placebo' group. As such, there was no data to analyze from these participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D and Omega-3 Fatty Acids | Vitamin D and Omega-3 Fatty Acid Placebo | Vitamin D Placebo and Omega-3 Fatty Acids | Vitamin D Placebo and Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 511 | 529 | 543 | 506
Participants | 4 | 6 | 6 | 6

ADVERSE EVENTS:
Time Frame: 4 years
Description: This ancillary study is not administering any treatments. All treatment monitoring occurred through the parent VITAL study (NCT01169259). The only adverse events obtained were in conjunction with results from laboratory samples collected for analysis at ~4 years
Arm/Group | Vitamin D and Omega-3 Fatty Acids | Vitamin D and Omega-3 Fatty Acid Placebo | Vitamin D Placebo and Omega-3 Fatty Acids | Vitamin D Placebo and Omega-3 Fatty Acids Placebo
All-Cause Mortality (participants affected / at risk) | 0/545 | 0/570 | 0/576 | 0/541
Serious Adverse Events (participants affected / at risk) | 0/545 | 0/570 | 0/576 | 0/541
Other Adverse Events (participants affected / at risk) | 4/545 | 6/570 | 6/576 | 6/541
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D and Omega-3 Fatty Acids (N=545) | Vitamin D and Omega-3 Fatty Acid Placebo (N=570) | Vitamin D Placebo and Omega-3 Fatty Acids (N=576) | Vitamin D Placebo and Omega-3 Fatty Acids Placebo (N=541)
Microalbuminuria (Renal and urinary disorders) | 4 | 6 | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT02757872/Prot_000.pdf